CLINICAL TRIAL: NCT03943550
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Phase Ib Study to Investigate the Safety, Tolerability, Pharmacokinetics, Preliminary Efficacy, and Pharmacodynamics of Subcutaneously Administered RO7049665 in Participants With Active Ulcerative Colitis
Brief Title: Double-Blinded, Placebo-Controlled Phase 1b Study for Safety, PK, Efficacy, PD of RO7049665 in Participants With Ulcerative Colitis (UC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to terminate study WP40161 was based on that treatment with RO7049665 showed trends in efficacy, however these data were below expectations and would not have supported superiority over standard of care.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: WP40161; 2017-004599-74 (EudraCT Number)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RO7049665 (Experimental): Participants will receive a subcutaneous (SC) dose of RO7049665 every 2 weeks for 4 doses.
  Interventions: Drug: RO7049665
- Placebo (Placebo Comparator): Participants will receive a SC dose of matching placebo every 2 weeks for 4 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RO7049665 — Multiple ascending doses of RO7049665 will be administered SC.
  Arms: RO7049665
Drug: Placebo — Matching placebo will be administered SC.
  Arms: Placebo

SUMMARY:
The principal aim of this study is to evaluate the safety and tolerability of RO7049665 in participants with active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with UC for at least 12 weeks prior to screening
* Screening colonoscopy for colorectal cancer conducted within the prior two years if a history of pancolitis with disease duration ≥ 8 years or history of left-sided colitis and disease duration ≥12 years
* Evidence of disease activity at time of screening
* Insufficient clinical response to standard of care (SOC) therapy or intolerance to SOC

Exclusion Criteria:

* Diagnosis of Crohn's disease or indeterminate colitis
* History of infection with hepatitis B, human immunodeficiency virus (HIV), active hepatitis C virus (HCV) infection, or other chronic infection
* Active infections requiring systemic therapy with antibiotic, antiviral or antifungal or febrile illness within 7 days before Day -1
* History of primary or acquired immunodeficiency
* Abnormal hematologic values
* Abnormal hepatic enzyme or hepatic function values

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Jacksonville Center for Clinical Research, Jacksonville, Florida, United States
- The Research Institute of Clinical Medicine, Tbilisi, Georgia
- Hungary (2):
  - Drug Research Centre Gyogyszervizsgalo Kozpontot Kft., Balatonfüred
  - SE ÁOK I. sz. Belgyógyászati Klinika, Budapest
- ARENSIA Phase 1 Unit- Spitalul Clinic Republican Location, Chisinau, Moldova
- Medical center of Yuriy Spizhenko LLC, Kapitanovka Village, KIEV Governorate, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 4 investigative centers in 4 countries Georgia, Hungary, Moldova, Ukraine from 13 May 2019 to 22 July 2021.
Pre-assignment Details: Participants with active ulcerative colitis (UC) were enrolled in the study.
Groups:
- Placebo: Participants received RO7049665 matching placebo, as subcutaneous (SC) injection, every 2 weeks for 4 doses up to Day 43 of the treatment period.
- RO7049665 3.5 mg: Participants received RO7049665, 3.5 milligrams (mg) as SC injection, every 2 weeks for 4 doses up to Day 43 of the treatment period.
- RO7049665 7.5 mg: Participants received RO7049665, 7.5 mg as SC injection, every 2 weeks for 4 doses up to Day 43 of the treatment period.
Period: Overall Study
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Started | 9 | 9 | 27
Completed | 9 | 8 | 23
Not Completed | 0 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 2
Not completed — Participant Moved Out of the Country | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Placebo: Participants received RO7049665 matching placebo, as SC injection, every 2 weeks for 4 doses up to Day 43 of the treatment period.
- RO7049665 3.5 mg: Participants received RO7049665, 3.5 mg as SC injection, every 2 weeks for 4 doses up to Day 43 of the treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg | Total
Number analyzed (Participants) | 9 | 9 | 27 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (17.5) | 35.1 (12.4) | 46.4 (11.8) | 43.3 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 13 | 20
  Male | 3 | 8 | 14 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 27 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 9 | 27 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE was defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity or is a congenital anomaly/birth defect. Severity of AEs were graded according to NCI CTCAE v4.0.
Time Frame: From baseline up to safety follow-up visit on Day 99
Population: Safety population included all participants randomized to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 9 | 27
Participants
  Number of participants with at least 1 AE | 4 | 6 | 24
  Number of participants with at least one SAE | 0 | 0 | 1

2. Secondary Outcome: Time to Maximum Concentration (Tmax) of RO7049665
Time Frame: Day 1 to Day 15 (predose) and Day 43 (post-dose)
Population: Pharmacokinetic (PK) analysis population included participants who had received active treatment. Number analyzed is the number of participants with evaluable data at specified timepoint.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 27
hour (h)
  Day 1-Day 15: Dose 1 | 12.00 [6.00 to 24.00] | 24.00 [6.00 to 72.08]
  Day 43: Dose 4: number analyzed (Participants) | 8 | 21
  Day 43: Dose 4 | 18.06 [12.00 to 72.57] | 24.00 [12.00 to 73.17]

3. Secondary Outcome: Maximum Serum Concentration Observed (Cmax) of RO7049665
Time Frame: Days 1 and 43: Pre-dose, 6 h and 12 h post-dose
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: nanograms per milliliters (ng/mL)
Groups:
- RO7049665 7.5mg: Participants received RO7049665, 7.5 mg as SC injection, every 2 weeks for 4 doses up to Day 43 of the treatment period.
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5mg
Number analyzed (Participants) | 9 | 27
nanograms per milliliters (ng/mL)
  Day 1: Dose 1 | 22.5 [8.59 to 63.7] | 47.6 [13.9 to 250]
  Day 43: Dose 4: number analyzed (Participants) | 8 | 21
  Day 43: Dose 4 | 38.7 [21.8 to 65.4] | 46.5 [20.2 to 109]

4. Secondary Outcome: Area Under the Serum Concentration-time Curve Extrapolated to Infinity (AUCinf) of RO7049665
Time Frame: Days 1 and 43: Pre-dose, 6 h and 12 h post-dose
Population: PK analysis population included participants who had received active treatment. Number analyzed is the number of participants with evaluable data at specified timepoint.
Measure: Geometric Mean (Full Range); unit: h*ng/mL
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 27
h*ng/mL
  Day 1: Dose 1 | 2030 [1020 to 3550] | 4520 [1780 to 15100]
  Day 43: Dose 4: number analyzed (Participants) | 8 | 21
  Day 43: Dose 4 | 3520 [1830 to 5740] | 4110 [2200 to 8240]

5. Secondary Outcome: Change From Baseline in the Endoscopy Subscore of the Mayo Clinic Score (MCS-ES)
Description: The Mayo Clinic Score (MCS) ranges from 0 to 12 and is a composite of 4 assessments, each rated from 0-3: stool frequency, rectal bleeding, endoscopy (i.e., centrally read MCS-ES) and Physician Global Assessment (PGA). Flexible sigmoidoscopy (or colonoscopy) was centrally read and scored using the MCS-ES scoring systems. The disease was considered as endoscopic normal or inactive if the MCS-ES (centrally read) was 0, mild (erythema, decreased vascular pattern) if MCS-ES was 1, moderate (marked erythema, absent vascular pattern, erosions) if MCS-ES was 2 and severe (spontaneous bleeding, ulceration) if MCS-ES was 3. The Endoscopy Subscore of the Mayo Score was modified so that a value of 1 did not include friability. A negative change from baseline indicates improvement.
Time Frame: Baseline, Days 29 and 57
Population: ITT population included all randomized participants. Number analyzed is the number of participants with evaluable data at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 9 | 27
score on a scale
  Baseline | 2.56 (0.53) | 2.44 (0.53) | 2.59 (0.50)
  Change from Baseline at Day 29: number analyzed (Participants) | 9 | 9 | 24
  Change from Baseline at Day 29 | -0.22 (0.83) | -0.22 (0.83) | -0.54 (0.98)
  Change from Baseline at Day 57: number analyzed (Participants) | 9 | 8 | 24
  Change from Baseline at Day 57 | -0.11 (0.93) | 0.00 (0.53) | -0.42 (0.72)

6. Secondary Outcome: Change From Baseline in the Ulcerative Colitis Endoscopic Index of Severity (UCEIS)
Description: Flexible sigmoidoscopy (or colonoscopy) were centrally read and scored using the UCEIS scoring systems. The UCEIS total score is a sum of 3 assessments: Bleeding (scored 0-3), Erosion and Ulcers (scored 0-3), and Vascular Pattern (scored 0-2). The total score ranges from 0-8, with higher score indicating more severe disease. A negative change from baseline indicates improvement.
Time Frame: Baseline, Days 29 and 57
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 9 | 27
score on a scale
  Baseline | 4.33 (1.12) | 4.00 (1.73) | 3.85 (0.86)
  Change from Baseline at Day 29: number analyzed (Participants) | 9 | 9 | 24
  Change from Baseline at Day 29 | -0.67 (1.32) | -0.22 (1.79) | -0.71 (1.52)
  Change from Baseline at Day 57: number analyzed (Participants) | 9 | 8 | 24
  Change from Baseline at Day 57 | -0.22 (1.56) | 0.63 (1.85) | -0.71 (1.33)

7. Secondary Outcome: Change From Baseline in Histology Score of Sigmoid Colon Biopsies Using Geboes Score (GS)
Description: Mucosal biopsies were obtained during flexible sigmoidoscopy from the most affected area 10 to 20 centimeters (cm) from the anal verge. Biopsies were assessed by standard histology for changes in the inflammatory activity as measured using GS. The GS is a stepwise grading system used for the evaluation of microscopic inflammation and histopathologic disease activity in UC. The microscopic appearance of the mucosa is categorized into 6 grades: Grade 0: architectural changes, Grade 1: chronic inflammatory infiltrate, Grade 2: lamina propria neutrophils and eosinophils, Grade 3: neutrophils in epithelium, Grade 4: crypt destruction and erosions or Grade 5: ulcerations, and each grade of the score is divided in 4 subcategories. A decrease of the Geboes grading system to Grades 0 or 1 would indicate mucosal healing.
Time Frame: Baseline, Days 29 and 57
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 9 | 26
score on a scale
  Baseline | 4.56 (0.88) | 3.22 (1.92) | 3.54 (2.04)
  Change from Baseline at Day 29: number analyzed (Participants) | 9 | 9 | 23
  Change from Baseline at Day 29 | -0.33 (1.22) | 0.78 (2.49) | -0.70 (1.11)
  Change from Baseline at Day 57: number analyzed (Participants) | 9 | 8 | 24
  Change from Baseline at Day 57 | -0.89 (1.90) | 0.88 (2.85) | -0.54 (1.82)

8. Secondary Outcome: Change From Baseline in Histology Score of Sigmoid Colon Biopsies Using Robarts Histology Index (RHI)
Description: Mucosal biopsies were obtained during flexible sigmoidoscopy from the most affected area 10 to 20 cm from the anal verge. Biopsies were assessed by standard histology for changes in the inflammatory activity as measured using RIH. The RHI is an evaluative index, derived from the Geboes score and is designed to be reproducible and responsive to clinically meaningful change in disease activity over time. The total RHI score ranges from 0 (no disease activity) to 33 (severe disease activity). A negative change from baseline indicates improvement.
Time Frame: Baseline, Days 29 and 57
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 9 | 26
score on a scale
  Baseline | 18.78 (7.19) | 11.44 (9.30) | 14.88 (10.90)
  Change from Baseline at Day 29: number analyzed (Participants) | 9 | 9 | 23
  Change from Baseline at Day 29 | -3.11 (8.52) | 3.89 (11.85) | -3.17 (7.36)
  Change from Baseline at Day 57: number analyzed (Participants) | 9 | 8 | 24
  Change from Baseline at Day 57 | -6.22 (8.91) | 5.38 (16.83) | -1.25 (8.90)

9. Secondary Outcome: Change From Baseline in Histology Score of Sigmoid Colon Biopsies Using Nancy Histology Index (NHI)
Description: Mucosal biopsies were obtained during flexible sigmoidoscopy from the most affected area 10 to 20 cm from the anal verge. Biopsies were assessed by standard histology for changes in the inflammatory activity as measured using NHI. NHI is a validated index for assessing histological disease activity in UC. It is composed of three histological items defining five grades of disease activity: absence of significant histological disease (Grade 0), chronic inflammatory infiltrate with no acute inflammatory infiltrate (Grade 1), mildly active disease (Grade 2), moderately active disease (Grade 3), and severely active disease (Grade 4). The presence of ulceration on the biopsy specimen corresponds to severely active disease (Grade 4). A decrease of the NHI grading system to Grades 0 or 1 would indicate improvement.
Time Frame: Baseline, Days 29 and 57
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 9 | 26
score on a scale
  Baseline | 3.11 (0.78) | 2.11 (1.45) | 2.42 (1.68)
  Change from Baseline at Day 29: number analyzed (Participants) | 9 | 9 | 23
  Change from Baseline at Day 29 | -0.56 (1.01) | 0.33 (1.94) | -0.57 (1.08)
  Change from Baseline at Day 57: number analyzed (Participants) | 9 | 8 | 24
  Change from Baseline at Day 57 | -0.78 (1.48) | 0.88 (2.42) | -0.25 (1.29)

10. Secondary Outcome: Percentage of Participants With Mayo Clinic Score (MCS) Clinical Response
Description: The MCS ranges from 0 to 12 and is a composite of 4 assessments: stool frequency, rectal bleeding, endoscopy (i.e., centrally read MCS-ES) and Physician Global Assessment (PGA). Each assessment was rated from 0-3, with higher score indicating more severe disease. Clinical response was defined as a decrease in the MCS of at least 3 points and at least 30% decrease from baseline.
Time Frame: Baseline, Days 29 and 57
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5mg
Number analyzed (Participants) | 9 | 9 | 27
percentage of participants
  Day 29: number analyzed (Participants) | 9 | 9 | 24
  Day 29 | 11.1 [0.28 to 48.25] | 33.3 [7.49 to 70.07] | 16.7 [4.74 to 37.38]
  Day 57: number analyzed (Participants) | 9 | 8 | 24
  Day 57 | 22.2 [2.81 to 60.01] | 50.0 [15.7 to 84.3] | 45.8 [25.55 to 67.18]

11. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs)
Description: ADA assays was used to detect anti-drug antibodies against RO7049665. Samples which were positive for anti-drug antibodies were further assessed using a neutralizing antibody assay. Participants were considered ADA positive if they were ADA negative at baseline but developed an ADA response following study drug administration (treatment-induced ADA response), or if they were ADA positive at baseline and the titer of one or more post-baseline samples was greater than the titer of the baseline sample by a scientifically reasonable margin such as at least 4-fold (treatment-enhanced ADA response).
Time Frame: Baseline; Post-dose on Days 8, 22, 57, 71 and 99; Pre-dose on Days 15, 29 and 43
Population: Immunogenicity population included all participants who had at least one pre-dose and one post-dose ADA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 9 | 27
Participants
  ADA Positive: Treatment-Induced ADA Response | 0 | 6 | 18
  ADA Positive: Treatment-Enhanced ADA Response | 0 | 0 | 2

12. Secondary Outcome: Change From Baseline in White Blood Cells (Tregs, Teffs)
Time Frame: Baseline; Pre-dose: Days 15, 29 and 43; Post-dose: Days 2, 6, 8, 10, 22, 36, 48, 50, 52, 57, 71
Population: Safety population included all participants randomized to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not. Number analyzed is the number of participants with evaluable data at specified timepoint.
Measure: Mean (Standard Deviation); unit: cells/µl
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 9 | 27
cells/µl
  CD4 Treg: Baseline: number analyzed (Participants) | 8 | 7 | 24
  CD4 Treg: Baseline | 37.25 (33.34) | 42.14 (25.07) | 51.21 (35.09)
  CD4 Treg: Change from Baseline at Day 2: number analyzed (Participants) | 6 | 6 | 17
  CD4 Treg: Change from Baseline at Day 2 | -2.83 (9.33) | -24.33 (19.51) | -25.65 (14.19)
  CD4 Treg: Change from Baseline at Day 6: number analyzed (Participants) | 6 | 5 | 19
  CD4 Treg: Change from Baseline at Day 6 | 12.17 (22.53) | 61.80 (31.22) | 87.37 (66.84)
  CD4 Treg: Change from Baseline at Day 8: number analyzed (Participants) | 7 | 6 | 22
  CD4 Treg: Change from Baseline at Day 8 | 3.00 (15.32) | 66.00 (68.26) | 169.34 (138.21)
  CD4 Treg: Change from Baseline at Day 10: number analyzed (Participants) | 4 | 5 | 18
  CD4 Treg: Change from Baseline at Day 10 | -8.25 (6.76) | 27.20 (18.99) | 137.81 (98.51)
  CD4 Treg: Change from Baseline at Day 15 (Pre-dose): number analyzed (Participants) | 5 | 7 | 22
  CD4 Treg: Change from Baseline at Day 15 (Pre-dose) | -3.80 (11.57) | 16.29 (28.42) | 37.73 (41.74)
  CD4 Treg: Change from Baseline at Day 22: number analyzed (Participants) | 6 | 7 | 21
  CD4 Treg: Change from Baseline at Day 22 | 5.17 (5.89) | 76.00 (70.04) | 186.45 (130.40)
  CD4 Treg: Change from Baseline at Day 29 (Pre-dose): number analyzed (Participants) | 8 | 7 | 19
  CD4 Treg: Change from Baseline at Day 29 (Pre-dose) | -3.75 (6.55) | 15.57 (18.74) | 27.66 (29.09)
  CD4 Treg: Change from Baseline at Day 36: number analyzed (Participants) | 7 | 5 | 19
  CD4 Treg: Change from Baseline at Day 36 | 4.57 (11.92) | 56.80 (57.37) | 110.61 (72.94)
  CD4 Treg: Change from Baseline at Day 43 (Pre-dose): number analyzed (Participants) | 6 | 5 | 16
  CD4 Treg: Change from Baseline at Day 43 (Pre-dose) | 4.00 (13.32) | 36.80 (26.12) | 33.22 (53.39)
  CD4 Treg: Change from Baseline at Day 48: number analyzed (Participants) | 7 | 6 | 13
  CD4 Treg: Change from Baseline at Day 48 | 2.71 (12.46) | 74.50 (48.63) | 149.96 (129.48)
  CD4 Treg: Change from Baseline at Day 50: number analyzed (Participants) | 7 | 5 | 19
  CD4 Treg: Change from Baseline at Day 50 | 5.43 (14.53) | 110.40 (57.33) | 115.79 (149.90)
  CD4 Treg: Change from Baseline at Day 52: number analyzed (Participants) | 4 | 5 | 11
  CD4 Treg: Change from Baseline at Day 52 | 1.63 (7.50) | 93.20 (39.16) | 81.64 (83.51)
  CD4 Treg: Change from Baseline at Day 57: number analyzed (Participants) | 7 | 5 | 19
  CD4 Treg: Change from Baseline at Day 57 | 0.71 (11.46) | 44.00 (28.47) | 35.08 (58.97)
  CD4 Treg: Change from Baseline at Day 71: number analyzed (Participants) | 8 | 6 | 17
  CD4 Treg: Change from Baseline at Day 71 | 5.38 (12.46) | 16.67 (42.32) | 14.50 (45.04)
  CD4 Teff: Baseline: number analyzed (Participants) | 9 | 9 | 25
  CD4 Teff: Baseline | 513.11 (249.55) | 707.72 (360.77) | 678.04 (211.81)
  CD4 Teff: Change from Baseline at Day 2: number analyzed (Participants) | 7 | 7 | 19
  CD4 Teff: Change from Baseline at Day 2 | 35.36 (166.81) | -164.07 (178.26) | -191.79 (175.75)
  CD4 Teff: Change from Baseline at Day 6: number analyzed (Participants) | 6 | 9 | 20
  CD4 Teff: Change from Baseline at Day 6 | 130.75 (183.96) | 101.17 (486.37) | 13.23 (161.24)
  CD4 Teff: Change from Baseline at Day 8: number analyzed (Participants) | 8 | 9 | 24
  CD4 Teff: Change from Baseline at Day 8 | 96.50 (152.39) | 148.17 (352.08) | 232.48 (237.40)
  CD4 Teff: Change from Baseline at Day 10: number analyzed (Participants) | 6 | 9 | 20
  CD4 Teff: Change from Baseline at Day 10 | 99.08 (271.08) | 117.06 (212.04) | 328.00 (375.95)
  CD4 Teff: Change from Baseline at Day 15 (Pre-dose): number analyzed (Participants) | 7 | 9 | 23
  CD4 Teff: Change from Baseline at Day 15 (Pre-dose) | 145.07 (226.10) | 89.06 (182.77) | 24.48 (234.22)
  CD4 Teff: Change from Baseline at Day 22: number analyzed (Participants) | 8 | 9 | 23
  CD4 Teff: Change from Baseline at Day 22 | 85.25 (140.67) | 117.17 (296.90) | 237.22 (284.96)
  CD4 Teff: Change from Baseline at Day 29 (Pre-dose): number analyzed (Participants) | 9 | 9 | 20
  CD4 Teff: Change from Baseline at Day 29 (Pre-dose) | 2.67 (189.20) | 21.50 (289.32) | -46.28 (165.72)
  CD4 Teff: Change from Baseline at Day 36: number analyzed (Participants) | 8 | 8 | 21
  CD4 Teff: Change from Baseline at Day 36 | 48.13 (174.33) | -22.38 (204.94) | 154.17 (198.56)
  CD4 Teff: Change from Baseline at Day 43 (Pre-dose): number analyzed (Participants) | 7 | 8 | 20
  CD4 Teff: Change from Baseline at Day 43 (Pre-dose) | 55.50 (174.27) | 96.69 (261.72) | 72.65 (193.91)
  CD4 Teff: Change from Baseline at Day 48: number analyzed (Participants) | 8 | 8 | 15
  CD4 Teff: Change from Baseline at Day 48 | 73.88 (166.61) | 128.31 (518.60) | 182.40 (287.99)
  CD4 Teff: Change from Baseline at Day 50: number analyzed (Participants) | 8 | 8 | 21
  CD4 Teff: Change from Baseline at Day 50 | 79.63 (210.91) | 220.56 (293.51) | 226.19 (274.34)
  CD4 Teff: Change from Baseline at Day 52: number analyzed (Participants) | 5 | 7 | 15
  CD4 Teff: Change from Baseline at Day 52 | 117.60 (160.56) | 199.64 (309.23) | 302.03 (282.02)
  CD4 Teff: Change from Baseline at Day 57: number analyzed (Participants) | 8 | 8 | 20
  CD4 Teff: Change from Baseline at Day 57 | 1.63 (154.15) | 202.56 (315.23) | 28.70 (194.94)
  CD4 Teff: Change from Baseline at Day 71: number analyzed (Participants) | 9 | 8 | 19
  CD4 Teff: Change from Baseline at Day 71 | 80.89 (138.90) | 142.81 (229.77) | -31.68 (158.78)
  CD8 Teff: Baseline: number analyzed (Participants) | 9 | 9 | 25
  CD8 Teff: Baseline | 178.22 (125.11) | 282.78 (226.36) | 272.40 (134.63)
  CD8 Teff: Change from Baseline at Day 2: number analyzed (Participants) | 7 | 7 | 19
  CD8 Teff: Change from Baseline at Day 2 | 15.57 (47.73) | -83.00 (109.30) | -43.87 (90.73)
  CD8 Teff: Change from Baseline at Day 6: number analyzed (Participants) | 6 | 9 | 20
  CD8 Teff: Change from Baseline at Day 6 | 63.08 (107.79) | 5.33 (242.60) | -16.23 (96.79)
  CD8 Teff: Change from Baseline at Day 8: number analyzed (Participants) | 8 | 9 | 24
  CD8 Teff: Change from Baseline at Day 8 | 27.38 (63.78) | 12.89 (159.82) | 67.40 (127.56)
  CD8 Teff: Change from Baseline at Day 10: number analyzed (Participants) | 6 | 9 | 20
  CD8 Teff: Change from Baseline at Day 10 | 24.83 (113.33) | 41.78 (125.23) | 115.35 (216.62)
  CD8 Teff: Change from Baseline at Day 15 (Pre-dose): number analyzed (Participants) | 7 | 9 | 23
  CD8 Teff: Change from Baseline at Day 15 (Pre-dose) | 56.21 (72.60) | -68.33 (119.93) | 8.00 (105.56)
  CD8 Teff: Change from Baseline at Day 22: number analyzed (Participants) | 8 | 9 | 23
  CD8 Teff: Change from Baseline at Day 22 | 31.25 (64.06) | -23.89 (247.21) | 68.52 (152.91)
  CD8 Teff: Change from Baseline at Day 29 (Pre-dose): number analyzed (Participants) | 9 | 9 | 20
  CD8 Teff: Change from Baseline at Day 29 (Pre-dose) | 5.67 (81.40) | -81.56 (170.89) | -27.85 (117.53)
  CD8 Teff: Change from Baseline at Day 36: number analyzed (Participants) | 8 | 8 | 21
  CD8 Teff: Change from Baseline at Day 36 | -9.00 (56.32) | -23.81 (72.26) | 94.21 (121.77)
  CD8 Teff: Change from Baseline at Day 43 (Pre-dose): number analyzed (Participants) | 7 | 8 | 20
  CD8 Teff: Change from Baseline at Day 43 (Pre-dose) | -0.29 (58.42) | 5.19 (100.23) | 21.15 (108.79)
  CD8 Teff: Change from Baseline at Day 48: number analyzed (Participants) | 8 | 8 | 15
  CD8 Teff: Change from Baseline at Day 48 | 11.00 (62.64) | 26.44 (213.36) | 63.07 (148.04)
  CD8 Teff: Change from Baseline at Day 50: number analyzed (Participants) | 8 | 8 | 21
  CD8 Teff: Change from Baseline at Day 50 | 18.38 (72.51) | 49.06 (153.58) | 83.10 (154.47)
  CD8 Teff: Change from Baseline at Day 52: number analyzed (Participants) | 5 | 7 | 15
  CD8 Teff: Change from Baseline at Day 52 | 50.60 (17.31) | 41.79 (143.04) | 105.47 (181.80)
  CD8 Teff: Change from Baseline at Day 57: number analyzed (Participants) | 8 | 8 | 20
  CD8 Teff: Change from Baseline at Day 57 | -16.50 (63.83) | 52.81 (200.84) | 25.33 (130.86)
  CD8 Teff: Change from Baseline at Day 71: number analyzed (Participants) | 9 | 8 | 19
  CD8 Teff: Change from Baseline at Day 71 | 17.89 (64.96) | 11.69 (114.91) | 21.82 (122.91)

13. Secondary Outcome: Change From Baseline in White Blood Cells (Natural Killer (NK) Cells)
Time Frame: Baseline; Pre-dose: Days 15, 29 and 43; Post-dose: Days 2, 6, 8, 10, 22, 36, 48, 50, 52, 57, 71
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: cells/µl
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 9 | 27
cells/µl
  Baseline | 146.44 (71.80) | 154.00 (102.99) | 227.24 (157.93)
  Change from Baseline at Day 2: number analyzed (Participants) | 8 | 9 | 24
  Change from Baseline at Day 2 | 2.31 (47.27) | 13.22 (59.30) | 34.56 (157.84)
  Change from Baseline at Day 6: number analyzed (Participants) | 8 | 9 | 26
  Change from Baseline at Day 6 | 86.88 (130.28) | 56.67 (114.71) | 57.77 (119.77)
  Change from Baseline at Day 8: number analyzed (Participants) | 8 | 9 | 26
  Change from Baseline at Day 8 | 26.44 (75.75) | 105.67 (72.36) | 73.90 (128.85)
  Change from Baseline at Day 10: number analyzed (Participants) | 8 | 9 | 24
  Change from Baseline at Day 10 | 53.94 (55.97) | 77.33 (125.77) | 119.31 (131.70)
  Change from Baseline at Day 15 (Pre-dose): number analyzed (Participants) | 8 | 9 | 27
  Change from Baseline at Day 15 (Pre-dose) | 4.44 (51.40) | 20.89 (45.83) | -25.35 (85.97)
  Change from Baseline at Day 22: number analyzed (Participants) | 8 | 9 | 26
  Change from Baseline at Day 22 | 26.19 (40.55) | 47.44 (84.33) | 93.81 (167.15)
  Change from Baseline at Day 29 (Pre-dose): number analyzed (Participants) | 9 | 9 | 22
  Change from Baseline at Day 29 (Pre-dose) | -6.78 (136.64) | -39.00 (52.92) | 40.84 (165.59)
  Change from Baseline at Day 36: number analyzed (Participants) | 8 | 9 | 24
  Change from Baseline at Day 36 | 14.44 (44.87) | 28.44 (32.84) | 75.46 (109.53)
  Change from Baseline at Day 43 (Pre-dose): number analyzed (Participants) | 8 | 8 | 23
  Change from Baseline at Day 43 (Pre-dose) | -2.44 (67.43) | -2.94 (37.03) | -5.72 (75.02)
  Change from Baseline at Day 48: number analyzed (Participants) | 9 | 8 | 23
  Change from Baseline at Day 48 | 42.89 (71.22) | 72.19 (33.30) | 109.65 (130.12)
  Change from Baseline at Day 50: number analyzed (Participants) | 8 | 8 | 24
  Change from Baseline at Day 50 | 31.88 (108.11) | 46.19 (65.72) | 97.58 (107.00)
  Change from Baseline at Day 52: number analyzed (Participants) | 9 | 8 | 21
  Change from Baseline at Day 52 | 48.33 (55.65) | 56.31 (60.30) | 111.38 (137.55)
  Change from Baseline at Day 57: number analyzed (Participants) | 8 | 8 | 23
  Change from Baseline at Day 57 | 28.69 (119.08) | 50.69 (74.56) | 30.52 (102.02)
  Change from Baseline at Day 71: number analyzed (Participants) | 9 | 8 | 21
  Change from Baseline at Day 71 | 47.44 (65.41) | 49.94 (39.55) | 35.19 (88.44)

14. Secondary Outcome: Change From Baseline in White Blood Cells (B Cells)
Time Frame: Baseline; Pre-dose: Days 15, 29 and 43; Post-dose: Days 2, 6, 8, 10, 22, 36, 48, 50, 52, 57, 71
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: cells/µl
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 9 | 27
cells/µl
  Baseline | 117.39 (51.86) | 149.39 (75.67) | 158.20 (76.23)
  Change from Baseline at Day 2: number analyzed (Participants) | 8 | 9 | 24
  Change from Baseline at Day 2 | -8.75 (26.26) | -30.06 (35.54) | -43.08 (36.06)
  Change from Baseline at Day 6: number analyzed (Participants) | 8 | 9 | 26
  Change from Baseline at Day 6 | 29.69 (53.88) | 27.94 (115.62) | -41.87 (47.32)
  Change from Baseline at Day 8: number analyzed (Participants) | 8 | 9 | 26
  Change from Baseline at Day 8 | 5.31 (31.10) | 29.17 (73.38) | 14.50 (39.33)
  Change from Baseline at Day 10: number analyzed (Participants) | 8 | 9 | 24
  Change from Baseline at Day 10 | 7.75 (24.33) | 37.72 (53.45) | 48.83 (48.94)
  Change from Baseline at Day 15 (Pre-dose): number analyzed (Participants) | 8 | 9 | 27
  Change from Baseline at Day 15 (Pre-dose) | 4.44 (34.11) | 30.61 (59.27) | 17.24 (46.26)
  Change from Baseline at Day 22: number analyzed (Participants) | 8 | 9 | 26
  Change from Baseline at Day 22 | 5.31 (28.01) | 18.06 (51.74) | 25.65 (52.69)
  Change from Baseline at Day 29 (Pre-dose): number analyzed (Participants) | 9 | 9 | 22
  Change from Baseline at Day 29 (Pre-dose) | -8.28 (35.09) | -5.06 (38.13) | -7.02 (33.59)
  Change from Baseline at Day 36: number analyzed (Participants) | 8 | 9 | 24
  Change from Baseline at Day 36 | -0.75 (28.83) | 17.50 (69.03) | 22.52 (39.02)
  Change from Baseline at Day 43 (Pre-dose): number analyzed (Participants) | 8 | 8 | 23
  Change from Baseline at Day 43 (Pre-dose) | 19.25 (51.24) | 23.13 (55.97) | 23.54 (47.44)
  Change from Baseline at Day 48: number analyzed (Participants) | 9 | 8 | 23
  Change from Baseline at Day 48 | 2.39 (25.68) | 22.88 (47.57) | 1.04 (40.30)
  Change from Baseline at Day 50: number analyzed (Participants) | 8 | 8 | 24
  Change from Baseline at Day 50 | 7.81 (37.53) | 28.00 (53.38) | 35.19 (62.64)
  Change from Baseline at Day 52: number analyzed (Participants) | 9 | 8 | 21
  Change from Baseline at Day 52 | 2.28 (31.15) | 20.63 (58.57) | 59.60 (53.87)
  Change from Baseline at Day 57: number analyzed (Participants) | 8 | 8 | 23
  Change from Baseline at Day 57 | -26.88 (23.22) | 24.13 (56.16) | 10.04 (60.22)
  Change from Baseline at Day 71: number analyzed (Participants) | 9 | 8 | 21
  Change from Baseline at Day 71 | -9.72 (16.36) | 4.38 (66.38) | 8.05 (52.65)

15. Secondary Outcome: Change From Baseline in Eosinophils
Time Frame: Baseline; Pre-dose: Days 15, 29 and 43; Post-dose: Days 2, 8, 22, 36, 57, 71 and follow-up visit on Day 99
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
Number analyzed (Participants) | 9 | 9 | 27
10^9/L
  Baseline | 0.177 (0.200) | 0.233 (0.275) | 0.204 (0.129)
  Change from Baseline at Day 2 | -0.014 (0.053) | 0.047 (0.088) | 0.047 (0.081)
  Change from Baseline at Day 8 | -0.009 (0.088) | 0.213 (0.141) | 0.387 (0.207)
  Change from Baseline at Day 15 (Pre-dose) | -0.010 (0.098) | 0.080 (0.170) | 0.283 (0.486)
  Change from Baseline at Day 22 | 0.008 (0.072) | 0.286 (0.214) | 1.373 (1.613)
  Change from Baseline at Day 29 (Pre-dose): number analyzed (Participants) | 9 | 9 | 24
  Change from Baseline at Day 29 (Pre-dose) | 0.021 (0.197) | 0.041 (0.199) | 0.318 (0.408)
  Change from Baseline at Day 36: number analyzed (Participants) | 9 | 9 | 24
  Change from Baseline at Day 36 | 0.014 (0.087) | 0.490 (0.340) | 1.234 (0.837)
  Change from Baseline at Day 43 (Pre-dose): number analyzed (Participants) | 9 | 8 | 24
  Change from Baseline at Day 43 (Pre-dose) | 0.000 (0.062) | 0.194 (0.210) | 0.386 (0.558)
  Change from Baseline at Day 57: number analyzed (Participants) | 9 | 8 | 24
  Change from Baseline at Day 57 | 0.022 (0.254) | 0.203 (0.232) | 0.378 (0.599)
  Change from Baseline at Day 71: number analyzed (Participants) | 9 | 8 | 24
  Change from Baseline at Day 71 | 0.031 (0.076) | 0.135 (0.155) | 0.085 (0.224)
  Change from Baseline at Day 99: number analyzed (Participants) | 9 | 8 | 23
  Change from Baseline at Day 99 | -0.022 (0.072) | 0.139 (0.286) | -0.019 (0.166)

ADVERSE EVENTS:
Time Frame: From baseline up to safety follow-up visit on Day 99
Description: Safety population included all participants randomized to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Arm/Group | Placebo | RO7049665 3.5 mg | RO7049665 7.5 mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 1/27
Other Adverse Events (participants affected / at risk) | 4/9 | 6/9 | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | RO7049665 3.5 mg (N=9) | RO7049665 7.5 mg (N=27)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | RO7049665 3.5 mg (N=9) | RO7049665 7.5 mg (N=27)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 13 (15)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 5 (17) | 18 (49)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT03943550/Prot_SAP_000.pdf